CLINICAL TRIAL: NCT00050037
Title: Cognitive Therapy Via CD-Rom for Binge-Eating Disorder
Brief Title: Cognitive Therapy for Binge-Eating Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Cynthia Bulik, PhD, Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21MH062053 (NIH); R21MH062053 (NIH); DSIR AT-AS
Record Dates: First submitted 2002-11-20; First posted 2002-11-21 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Obesity; Eating Disorders
MeSH Terms: conditions — Obesity; Feeding and Eating Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CD-ROM based CBT (Experimental): Group is given a copy of the CD-ROM program to complete at home over 10 weeks. At the end of each week, these patients upload and transmit their encrypted tracking data to the research coordinator. At the end of the treatment, participants who have not improved are offered a course of traditional manual-based group therapy, follow-up in an ongoing maintenance group in an eating disorders program, or an alternative treatment.
  Interventions: Procedure: CBT
- Standard Group CBT (Active Comparator): Group undergoes standard group CBT. Therapy is administered over 10 weeks in five 90-minute sessions. The key topics are similar to those covered in the CD-ROM group: psychoeducation, developing a personal profile, standardizing meal times, recognizing emotional eating, increasing daily activity, learning the language of CBT, identifying automatic thoughts, restructuring thoughts, identifying cues and consequences, chaining, "surfing the urge," and preventing relapses. Therapy sessions include a didactic section followed by group interaction and discussion. All group sessions are audiotaped and monitored.
  Interventions: Procedure: CBT
- Waiting List (No Intervention): Participants in the wait list control group undergo an initial assessment but receive no active intervention for 10 weeks. After 10 weeks, these patients undergo post-treatment assessment and are offered the opportunity to either enter group treatment in an eating disorders program or enter other appropriate treatment. Three-month follow-up data are not collected from these individuals.

INTERVENTIONS:
Procedure: CBT
  Other Names: Cognitive Behavioral Therapy
  Arms: CD-ROM based CBT; Standard Group CBT

SUMMARY:
The purpose of this study is to compare the efficacy of a CD-ROM-based cognitive-behavioral therapy (CBT) to traditional manual-based group therapy for obese individuals with binge-eating disorder (BED) and other unhealthy eating behaviors. A second goal is to encourage a healthy lifestyle in patients with BED.

DETAILED DESCRIPTION:
Although eating and weight-related disorders are treatable, most afflicted individuals never receive proper treatment.

CD-ROM-based CBT may be an efficacious and cost-effective intervention, a useful adjunct to traditional psychotherapy, or an introductory step to treatment which familiarizes patients with the principles and techniques of CBT and increases their comfort and motivation to seek additional help.

Potential participants undergo a brief telephone screening to ensure their understanding of the study. Individuals who meet preliminary criteria are then scheduled for an initial assessment.

Patients are randomized to 1 of 3 groups. One group is given a copy of the CD-ROM program to complete at home over 10 weeks. At the end of each week, these patients upload and transmit their encrypted tracking data to the research coordinator. At the end of the treatment, participants who have not improved are offered a course of traditional manual-based group therapy, follow-up in an ongoing maintenance group in an eating disorders program, or an alternative treatment.

A second group undergoes standard group CBT. Therapy is administered over 10 weeks in five 90-minute sessions. The key topics are similar to those covered in the CD-ROM group: psychoeducation, developing a personal profile, standardizing meal times, recognizing emotional eating, increasing daily activity, learning the language of CBT, identifying automatic thoughts, restructuring thoughts, identifying cues and consequences, chaining, "surfing the urge," and preventing relapses. Therapy sessions include a didactic section followed by group interaction and discussion. All group sessions are audiotaped and monitored.

Participants in the wait list control group undergo an initial assessment but receive no active intervention for 10 weeks. After 10 weeks, these patients undergo post-treatment assessment and are offered the opportunity to either enter group treatment in an eating disorders program or enter other appropriate treatment. Three-month follow-up data are not collected from these individuals.

Assessments occur at study start, at the end of treatment, and at a 3-month follow-up. Assessments include height and weight measurements and measurements of changes in exercise- and nonexercise-related activity. All participants are given tests and interviews to assess eating disorder symptoms, depression, psychoactive substance abuse and dependence, and functioning. Patients complete self-report questionnaires to assess their cognitive restraint, hunger, disinhibition, strength of urges to binge, and degree of confidence in their ability to resist a binge. Patients also rate the suitability of treatment both prior to and following completion of the intervention.

ELIGIBILITY:
Inclusion criteria:

* Binge-eating disorder (binging an average of once per week for 6 months)
* Body mass index of 30 or more
* Regular access to an IBM-compatible computer

Exclusion Criteria:

* Patients currently taking psychoactive medication will not be excluded provided their unhealthy eating behaviors have remained stable during treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2001-04; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States